CLINICAL TRIAL: NCT05585593
Title: Registry and Biobank for Patients With Hypoparathyroidism Wuerzburg
Brief Title: Registry for Hypoparathyroidism Wuerzburg
Status: Recruiting | Type: Observational
Sponsor: University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Stefanie Hahner, Prof. Dr., University of Wuerzburg
Other Study IDs: RESHOW
Record Dates: First submitted 2022-10-11; First posted 2022-10-19 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Comorbidities and Coexisting Conditions; Morality; Hypocalcemia; Hypercalcemia; Quality of Life
MeSH Terms: conditions — Hypocalcemia; Hypercalcemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Long-term conventional treatment of chronic hypoparathyroidism does not fully restore calcium homeostasis leading to increased morbidity, emergency events and reduced subjective health status. To further investigate general morbidity, hypocalcemic events, subjective and daily life performance in patients with chronic hypoparathyroidism a standardized interview as well as blood sampling and examinations such as echocardiography and renal ultrasound are performed.

DETAILED DESCRIPTION:
Design:

In a longitudinal prospective trial the comorbidities, mortality, hypocalcemic and hypercalcemic events and quality of life in patients with chronic hypoparathyroidism will be evaluated by a standardized interview, blood sampling and further examinations such as echocardiography and renal ultrasound.

Patients:

Patients will be recruited out of the patient population of the University Hospital Wuerzburg.

Statistical Analysis:

Documentation and analysis will be performed at the Department of Medicine I, Endocrine and Diabetes Unit, University of Würzburg, Germany. Data will be documented after pseudonymisation in a data base. For further analysis data will be compared to sex- and age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* age of 18
* chronic hypoparathyroidism (>12 months) under established therapy or chronic pseudohypoparathyroidism (>12 months) under established therapy
* written informed consent

Exclusion Criteria:

* age <18 years
* no detailed documentation of hypo- or pseudohypoparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic hypo- and pseudohypoparathyroidism
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Comorbidites | 15 years
  Comorbidities such as renal diseases, cardiovascular disease, psychiatric diseases under treatment
Subjective health status | 15 years
  Assessment of the subjective health status by standardized quality of life (QoL) questionnaires (e.g. short form-36, Patient Health Questionnaire 28)

SECONDARY OUTCOMES:
Hypocalcemic and hypercalcemic events | 15 years
  documentation of frequency of hypocalcemia under standard treatment
Mortality | 15 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Endocrinology and Diabetology, Dept. of Medicine I, University Hospital Wuerzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilezikian JP. Hypoparathyroidism. J Clin Endocrinol Metab. 2020 Jun 1;105(6):1722-36. doi: 10.1210/clinem/dgaa113. PMID 32322899
- [Background] Khan AA, AbuAlrob H, Punthakee Z, Shrayyef M, Werfalli RE, Kassem HA, Braga M, Millar A, Hussain S, Iqbal S, Khan T, Paul T, Van Uum S, Young JEM. Canadian national hypoparathyroidism registry: an overview of hypoparathyroidism in Canada. Endocrine. 2021 May;72(2):553-561. doi: 10.1007/s12020-021-02629-w. Epub 2021 Mar 2. PMID 33655415
- [Background] Underbjerg L, Sikjaer T, Mosekilde L, Rejnmark L. Cardiovascular and renal complications to postsurgical hypoparathyroidism: a Danish nationwide controlled historic follow-up study. J Bone Miner Res. 2013 Nov;28(11):2277-85. doi: 10.1002/jbmr.1979. PMID 23661265
- [Derived] Fuss CT, Gronemeyer K, Hermes F, Dorr M, Schmid B, Morbach C, Schmidbauer L, Schlegel N, Fassnacht M, Koschker AC, Nordbeck P, Hannemann A, Hahner S. Cardiovascular status in chronic hypoparathyroidism: a systematic cross-sectional assessment in 168 patients. Eur J Endocrinol. 2025 Mar 27;192(4):373-384. doi: 10.1093/ejendo/lvaf023. PMID 40172208
- [Derived] Gronemeyer K, Fuss CT, Hermes F, Plass A, Koschker AC, Hannemann A, Volzke H, Hahner S. Renal complications in chronic hypoparathyroidism - a systematic cross-sectional assessment. Front Endocrinol (Lausanne). 2023 Nov 2;14:1244647. doi: 10.3389/fendo.2023.1244647. eCollection 2023. PMID 38027217